CLINICAL TRIAL: NCT06529159
Title: H. Pylori Eradication With Argon Plasma During Endoscopy (HEAPE)
Brief Title: H. Pylori Eradication With Argon Plasma During Endoscopy
Acronym: HEAPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher C. Thompson, MD, MSc (Other)
Collaborators: Erbe Elektromedizin GmbH (Industry)
Responsible Party: Sponsor-Investigator, Christopher C. Thompson, MD, MSc, Director of Endoscopy, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024P002031
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Helicobacter Pylori Infection; Helicobacter Pylori; Helicobacter Pylori Gastrointestinal Tract Infection; H. Pylori Infection; H. Pylori Gastrointestinal Disease
Keywords: Urea Breath Test; Argon Plasma Coagulation (APC); Endoscopy; Plasma Activated Liquid (PAL); Plasma Medicine
MeSH Terms: interventions — Organization and Administration

STUDY DESIGN:
Intervention Model Description: Two-arm, randomized, pilot, single-center, prospective clinical study
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HEAPE direct (Active Comparator): This modality is the direct generation of PAL in the stomach. The stomach is filled with sodium chloride solution which is then treated with APC. With HEAPE direct a potential decrease of reactive species is avoided, as the treatment happens directly at the intended location in the H. pylori infected stomach.
  Interventions: Procedure: HEAPE
- Pre-HEAPE (Active Comparator): This modality features the treatment of sodium chloride with APC outside of the patient in a sterile container. After the APC treatment, the generated PAL is administered into the stomach with a syringe through the working channel of the endoscope. Pre-HEAPE allows an easier handling of the APC probe as the treatment of the sodium chloride solution can be done without an endoscope.
  Interventions: Procedure: Pre-HEAPE

INTERVENTIONS:
Procedure: HEAPE — The stomach is filled with sodium chloride solution which is then treated with APC to activate it into an antibacterial solution.
  Other Names: Endoscopic APC Treatment in vivo
  Arms: HEAPE direct
Procedure: Pre-HEAPE — Plasma activated sodium chloride solution (prepared outside of the body) is administered into the patients stomach through an endoscope channel using a syringe.
  Other Names: Plasma Activated Liquid (PAL) Administration
  Arms: Pre-HEAPE

SUMMARY:
The objective of the study is to investigate the efficacy and safety of an argon plasma-based therapy - HEAPE - in treating H. pylori infections during endoscopic procedures. By filling the stomach with sodium chloride solution that is treated with APC (PAL), the Investigators hypothesize a significant reduction in H. pylori. The use of PAL instead of direct application of APC allows for a broader and more homogeneous application throughout the stomach and a faster procedure time, as the fluid bypasses the thermal effects typically associated with higher electrical power settings and focuses on the bactericidal action of PAL. It is a procedure that does not involve thermal ablation of the stomach lining. Thus, side effects should be expected to be as low as possible.

Two different PAL generation modalities will be compared in this study:

1. HEAPE direct: This modality is the direct generation of PAL in the stomach. The stomach is filled with sodium chloride solution which is then treated with APC. With HEAPE direct a potential decrease of reactive species is avoided, as the treatment happens directly at the intended location in the H. pylori infected stomach.
2. Pre-HEAPE: This modality features the treatment of sodium chloride with APC outside of the patient in a sterile container. After the APC treatment, the generated PAL is administered into the stomach with a syringe through the working channel of the endoscope. Pre-HEAPE allows an easier handling of the APC probe as the treatment of the sodium chloride solution can be done without an endoscope.

To evaluate the immediate effect of this novel treatment approach the metabolic activity of H. pylori will be assessed using a urea breath test (UBT) before and after treatment. A reduction in H. pylori levels can be detected by a reduction in urease activity in the breath test.

After the HEAPE procedure, patients are treated with antibiotics (best practice) as they would be under normal circumstances. Four weeks after treatment, another UBT is performed to determine if H. pylori has been eradicated or if additional antibiotic treatment is indicated.

This two-arm, randomized, pilot, single-center, prospective clinical study is designed to evaluate the safety, tolerability and proof of concept that PAL has the ability to eradicate or reduce the bacterial load of H. pylori in humans.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) is a prevalent bacterial infection that colonizes the gastric mucosa, affecting approximately 50% of the global population. Classified by the WHO as a class 1 carcinogen in 1994 and further supported by extensive evidence, H. pylori is recognized as a leading cause of ulcers and a significant risk factor for the development of gastric cancer. Despite a slight decline in the prevalence of H. pylori infection in developed countries, the absolute number of infected individuals in the U.S. remains alarmingly high at approximately 36% of the U.S. population. Gastric cancer, associated with H. pylori infection, continues to be a major health concern worldwide, accounting for over 1.1 million new cases and approximately 770,000 deaths each year. The causal link between H. pylori infection and nearly 90% of gastric cancer cases underscores the critical importance of effective eradication strategies.

Current treatments for H. pylori infection, which typically consist of triple or quadruple therapy combining two or three antibiotics with proton pump inhibitors (PPIs), are successful in approximately 80% of cases. This leaves a significant proportion of cases unresolved. In addition, the emergence of multidrug-resistant H. pylori strains, particularly those resistant to clarithromycin and quinolones, challenges these conventional approaches. The broader issue of increasing antibiotic resistance, leads to a reliance on back-up antibiotics for cases where standard treatments fail. A sharp decline of eradication rates during the last decade, underscores the need for alternative therapeutic strategies. A recent study estimated the total cost of H. pylori treatment failure to be over $5.3 billion in the U.S., primarily due to hospitalizations, medications, and outpatient visits for complications such as peptic ulcer disease and non-cardia gastric cancer. Research into treatments beyond antibiotics is needed to address the growing risk of resistance and to ensure sustainable, effective solutions for H. pylori infection.

The field of plasma medicine, particularly through the use of Argon Plasma Coagulation (APC), offers promising new avenues for addressing this challenge. APC, a technology with over 30 years of clinical safety and efficacy, has been utilized for bleeding management, ablation of cancerous tissues, and precise treatments in sensitive areas. More recently, it has shown good efficacy in the treatment of cervical intraepithelial lesions (CIN) at lower power levels with no visible macroscopic thermal effect. Recent advancements in plasma medicine have highlighted the antibacterial properties of physical plasma. It has demonstrated remarkable efficacy in wound healing by effectively eradicating bacterial infections, including those resistant to antibiotics. The effect of non-thermal plasma treatment is based on the high energy and voltage of the plasma, which generates reactive oxygen and nitrogen species (RONS), an electric field that can cause electroporative effects, and UV light emitted in the plasma.

These effects are present when plasma is applied directly to the site of action, but also when a liquid medium such as sodium chloride solution is used as a buffer substance. This concept of indirect plasma treatment is often referred to as Plasma Activated Liquid (PAL). In proprietary preclinical studies, PAL generated with APC probes using forced APC Effect 8 has been shown to achieve a 5-log reduction in H. pylori (SK225) after 15 minutes incubation. In a multidrug resistant E. coli 4MRGN stain (VC8874), a 6-log reduction was achieved after 15 minutes incubation.

This demonstrates that PAL harnesses the antimicrobial properties of plasma in a non-thermal, liquid-based approach. This innovative approach allows the effects of plasma to be applied to large surface areas, such as the gastric mucosa, offering a potentially effective treatment for H. pylori infection without the drawbacks associated with antibiotic resistance. The established safety record of APC and the common use of liquids as irrigation or injection solutions in endoscopy provide a solid foundation for its potential applications in the treatment of H. pylori infection.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 years or older
2. Confirmed untreated H. pylori infection
3. Able to understand and sign informed consent
4. Available to return for all routine follow-up study visits
5. Patients should have upper endoscopy scheduled according to latest guidelines, e.g., as a part of their diagnostic work-up of HP positive test, regardless of their decision to participate in the study.

Exclusion Criteria:

1. Patients actively undergoing H.pylori eradication therapy treatment with antibiotics or proton pump inhibitors (PPIs) two weeks prior to the HEAPE procedure.
2. Pregnancy or puerperium
3. Severe cardiopulmonary disease or a history of coronary artery disease (including myocardial infarction within the past 6 months, poorly controlled hypertension, required use of NSAIDs)
4. Lactation
5. An inability to provide informed consent
6. Any other condition which the investigator may deem as an impediment to compliance or hinder completion of the proposed study.
7. Hernias / aspiration risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in H. pylori load from baseline to 2 hours after treatment using Urea Breath Test | Baseline, 2 hours post-treatment
  Change in measurement H. pylori metabolic activity using the Urea Breath Test (UBT) 1 (+2/-0) day before and 2 (+18/-0) hours after treatment

SECONDARY OUTCOMES:
Eradication of H. pylori load from 2 hours after treatment to 4 weeks after treatment using Urea Breath Test | 2 hours post-treatment, 4 weeks post-treatment
  H. pylori eradication (negative UBT) directly after the HEAPE treatment (timepoint 1) and 4 (+2/-0) weeks after HEAPE treatment (timepoint 2)
Comparison of H. pylori eradication rate between HEAPE + standard of care antibiotic treatment vs standard of care treatment (antibiotics) alone (historical data) | 4 weeks
  Comparison of eradication rates at 4 weeks between patients treated with HEAPE + antibiotics vs. published literature using UBT values
Comparison of reduction in H. pylori load measured by UBT HEAPE vs. Pre-HEAPE treatment arms from baseline to 2 hours post-treatment | Baseline, 2 hours post-treatment
  Comparison of the reduction in H. pylori load, as measured by Urea Breath Test (UBT), 2 (+18/-0) hours after treatment between the HEAPE direct modality and the Pre-HEAPE modality
Comparison of H. pylori load measured by UBT HEAPE vs. Pre-HEAPE treatment arms from baseline to 4 weeks post-treatment | Baseline, 4 weeks post-treatment
  Comparison of the reduction in H. pylori load, as measured by Urea Breath Test (UBT), 4 weeks after treatment between the HEAPE direct modality and the Pre-HEAPE modality
Change in dyspepsia symptoms from baseline via patient self-report of symptoms | Baseline, 4 weeks
  Change in patient self-report of dyspepsia symptoms from baseline up to 4 weeks post-treatment
Change in epigastric pain level from baseline via patient self-report of symptoms using the Abdominal Pain Index | Baseline, 4 weeks
  Change in patient self-report of epigastric pain level from baseline up to 4 weeks post-treatment using Abdominal Pain Index (from no pain (0) to the most pain possible (10)).
Change in quality of life score from baseline using the 12 item Short Form Survey (SF-12) | Baseline, 4 weeks
  Comparison of quality of life scores from baseline to 4 weeks post-treatment using the SF-12 scoring system. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning. A score of 50 or less has been recommended as a cut-off to determine a physical condition in the Physical Health Composite Score (PCS) section; while a score of 42 or less may be indicative of 'clinical depression' Mental Health Composite Score (MCS) section.
Adverse Events intra-procedural and post-treatment | Intra-procedure, 2 hours post-treatment, 4 weeks post-treatment
  Presence of adverse events that develop post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C Thompson, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared on a case by case basis with an Institutional data transfer agreement in place.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 12 months after publication
Access Criteria: IPD requests should be made directly to the PI who will determine feasibility of the request. Institutional data transfer agreement will need to be executed to share data.

REFERENCES:
- [Background] Hooi JKY, Lai WY, Ng WK, Suen MMY, Underwood FE, Tanyingoh D, Malfertheiner P, Graham DY, Wong VWS, Wu JCY, Chan FKL, Sung JJY, Kaplan GG, Ng SC. Global Prevalence of Helicobacter pylori Infection: Systematic Review and Meta-Analysis. Gastroenterology. 2017 Aug;153(2):420-429. doi: 10.1053/j.gastro.2017.04.022. Epub 2017 Apr 27. PMID 28456631
- [Background] Wang C, Yuan Y, Hunt RH. The association between Helicobacter pylori infection and early gastric cancer: a meta-analysis. Am J Gastroenterol. 2007 Aug;102(8):1789-98. doi: 10.1111/j.1572-0241.2007.01335.x. Epub 2007 May 23. PMID 17521398
- [Background] Mrochen DM, Miebach L, Skowski H, Bansemer R, Drechsler CA, Hofmanna U, Hein M, Mamat U, Gerling T, Schaible U, von Woedtke T, Bekeschus S. Toxicity and virucidal activity of a neon-driven micro plasma jet on eukaryotic cells and a coronavirus. Free Radic Biol Med. 2022 Oct;191:105-118. doi: 10.1016/j.freeradbiomed.2022.08.026. Epub 2022 Aug 28. PMID 36041652
- [Background] Liou JM, Malfertheiner P, Lee YC, Sheu BS, Sugano K, Cheng HC, Yeoh KG, Hsu PI, Goh KL, Mahachai V, Gotoda T, Chang WL, Chen MJ, Chiang TH, Chen CC, Wu CY, Leow AH, Wu JY, Wu DC, Hong TC, Lu H, Yamaoka Y, Megraud F, Chan FKL, Sung JJ, Lin JT, Graham DY, Wu MS, El-Omar EM; Asian Pacific Alliance on Helicobacter and Microbiota (APAHAM). Screening and eradication of Helicobacter pylori for gastric cancer prevention: the Taipei global consensus. Gut. 2020 Dec;69(12):2093-2112. doi: 10.1136/gutjnl-2020-322368. Epub 2020 Oct 1. PMID 33004546
- [Background] Cavaleiro-Pinto M, Peleteiro B, Lunet N, Barros H. Helicobacter pylori infection and gastric cardia cancer: systematic review and meta-analysis. Cancer Causes Control. 2011 Mar;22(3):375-87. doi: 10.1007/s10552-010-9707-2. Epub 2010 Dec 24. PMID 21184266
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Atherton J, Axon AT, Bazzoli F, Gensini GF, Gisbert JP, Graham DY, Rokkas T, El-Omar EM, Kuipers EJ; European Helicobacter Study Group. Management of Helicobacter pylori infection--the Maastricht IV/ Florence Consensus Report. Gut. 2012 May;61(5):646-64. doi: 10.1136/gutjnl-2012-302084. PMID 22491499
- [Background] Argueta EA, Alsamman MA, Moss SF, D'Agata EMC. Impact of Antimicrobial Resistance Rates on Eradication of Helicobacter pylori in a US Population. Gastroenterology. 2021 May;160(6):2181-2183.e1. doi: 10.1053/j.gastro.2021.02.014. Epub 2021 Feb 9. No abstract available. PMID 33577874
- [Background] Shiota S, Reddy R, Alsarraj A, El-Serag HB, Graham DY. Antibiotic Resistance of Helicobacter pylori Among Male United States Veterans. Clin Gastroenterol Hepatol. 2015 Sep;13(9):1616-24. doi: 10.1016/j.cgh.2015.02.005. Epub 2015 Feb 11. PMID 25681693
- [Background] Megraud F, Graham DY, Howden CW, Trevino E, Weissfeld A, Hunt B, Smith N, Leifke E, Chey WD. Rates of Antimicrobial Resistance in Helicobacter pylori Isolates From Clinical Trial Patients Across the US and Europe. Am J Gastroenterol. 2023 Feb 1;118(2):269-275. doi: 10.14309/ajg.0000000000002045. Epub 2022 Sep 30. PMID 36191284
- [Background] Shah S, Hubscher E, Pelletier C, Jacob R, Vinals L, Yadlapati R. Helicobacter pylori infection treatment in the United States: clinical consequences and costs of eradication treatment failure. Expert Rev Gastroenterol Hepatol. 2022 Apr;16(4):341-357. doi: 10.1080/17474124.2022.2056015. Epub 2022 Apr 1. PMID 35315732
- [Background] Zenker M. Argon plasma coagulation. GMS Krankenhhyg Interdiszip. 2008 Nov 3;3(1):Doc15. PMID 20204117
- [Background] Eickhoff A, Jakobs R, Schilling D, Hartmann D, Weickert U, Enderle MD, Eickhoff JC, Riemann JF. Prospective nonrandomized comparison of two modes of argon beamer (APC) tumor desobstruction: effectiveness of the new pulsed APC versus forced APC. Endoscopy. 2007 Jul;39(7):637-42. doi: 10.1055/s-2007-966571. PMID 17611919
- [Background] Kwan V, Bourke MJ, Williams SJ, Gillespie PE, Murray MA, Kaffes AJ, Henriquez MS, Chan RO. Argon plasma coagulation in the management of symptomatic gastrointestinal vascular lesions: experience in 100 consecutive patients with long-term follow-up. Am J Gastroenterol. 2006 Jan;101(1):58-63. doi: 10.1111/j.1572-0241.2006.00370.x. PMID 16405534
- [Background] Vargo JJ. Clinical applications of the argon plasma coagulator. Gastrointest Endosc. 2004 Jan;59(1):81-8. doi: 10.1016/s0016-5107(03)02296-x. No abstract available. PMID 14722558
- [Background] Grund KE, Straub T, Farin G. New haemostatic techniques: argon plasma coagulation. Baillieres Best Pract Res Clin Gastroenterol. 1999 Apr;13(1):67-84. doi: 10.1053/bega.1999.0009. PMID 11030635
- [Background] Grund KE, Zindel C, Farin G. [Argon plasma coagulation through a flexible endoscope. Evaluation of a new therapeutic method after 1606 uses]. Dtsch Med Wochenschr. 1997 Apr 4;122(14):432-8. doi: 10.1055/s-2008-1047634. German. PMID 9138921
- [Background] Grund KE, Storek D, Farin G. Endoscopic argon plasma coagulation (APC) first clinical experiences in flexible endoscopy. Endosc Surg Allied Technol. 1994 Feb;2(1):42-6. PMID 8081915
- [Background] Weiss M, Arnholdt M, Hissnauer A, Fischer I, Schonfisch B, Andress J, Gerstner S, Dannehl D, Bosmuller H, Staebler A, Brucker SY, Henes M. Tissue-preserving treatment with non-invasive physical plasma of cervical intraepithelial neoplasia-a prospective controlled clinical trial. Front Med (Lausanne). 2023 Aug 15;10:1242732. doi: 10.3389/fmed.2023.1242732. eCollection 2023. PMID 37654659
- [Background] Marzi J, Stope MB, Henes M, Koch A, Wenzel T, Holl M, Layland SL, Neis F, Bosmuller H, Ruoff F, Templin M, Kramer B, Staebler A, Barz J, Carvajal Berrio DA, Enderle M, Loskill PM, Brucker SY, Schenke-Layland K, Weiss M. Noninvasive Physical Plasma as Innovative and Tissue-Preserving Therapy for Women Positive for Cervical Intraepithelial Neoplasia. Cancers (Basel). 2022 Apr 12;14(8):1933. doi: 10.3390/cancers14081933. PMID 35454839
- [Background] Han Q, He ZY, Chongshan Z, Wen X, Ni YY. The optimization of plasma activated water (PAW) generation and the inactivation mechanism of PAW on Escherichia coli. Journal of Food Processing and Preservation. 2022;46(11):1-12.
- [Background] Traylor MJ, Pavlovich MJ, Karim S et al. Long-term antibacterial efficacy of air plasma-activated water. Plasma Sources Sci. Technol. 2011; 44: 472001
- [Background] Chen TP, Liang J, Su TL. Plasma-activated water: antibacterial activity and artifacts? Environ Sci Pollut Res Int. 2018 Sep;25(27):26699-26706. doi: 10.1007/s11356-017-9169-0. Epub 2017 May 24. PMID 28540555
- [Background] Schmidt M, Hahn V, Altrock B et al. Plasma-Activation of Larger Liquid Volumes by an Inductively-Limited Discharge for Antimicrobial Purposes. Applied Sciences 2019; 9: 2150
- [Background] Ma M, Zhang Y, Lv Y et al. The key reactive species in the bactericidal process of plasma activated water. Journal of Applied Physics 2020; 53:185207
- [Background] Mai-Prochnow A, Zhou R, Zhang T, Ostrikov KK, Mugunthan S, Rice SA, Cullen PJ. Interactions of plasma-activated water with biofilms: inactivation, dispersal effects and mechanisms of action. NPJ Biofilms Microbiomes. 2021 Jan 27;7(1):11. doi: 10.1038/s41522-020-00180-6. PMID 33504802
- [Background] Wang L, Xia C, Guo Y, Yang C, Cheng C, Zhao J, Yang X, Cao Z. Bactericidal efficacy of cold atmospheric plasma treatment against multidrug-resistant Pseudomonas aeruginosa. Future Microbiol. 2020 Jan;15:115-125. doi: 10.2217/fmb-2019-0265. Epub 2020 Jan 28. PMID 31989838
- [Background] Yang L, Niyazi G, Qi Y, Yao Z, Huang L, Wang Z, Guo L, Liu D. Plasma-Activated Saline Promotes Antibiotic Treatment of Systemic Methicillin-Resistant Staphylococcus aureus Infection. Antibiotics (Basel). 2021 Aug 22;10(8):1018. doi: 10.3390/antibiotics10081018. PMID 34439068
- [Background] Adamovich I, Agarwal S, Ahedo E et al. The 2022 Plasma Roadmap: low temperature plasma science and technology. Plasma Sources Sci. Technol. 2022; 55: 373001
- [Background] Wang Z, Qi Y, Guo L et al. The bactericidal effects of plasma-activated saline prepared by the combination of surface discharge plasma and plasma jet. Plasma Sources Sci. Technol. 2021; 54: 385202
- [Background] Zhao Y-M, Ojha S, Burgess CM et al. Inactivation efficacy of plasma-activated water: influence of plasma treatment time, exposure time and bacterial species. Int. J. Food Sci. Technol. 2021; 56: 721-732